CLINICAL TRIAL: NCT00403117
Title: Opioid Antagonism Enhances Marijuana's Effects in Heavy Marijuana Smokers
Brief Title: Effects of a Range of Naltrexone Doses in Combination With Smoked Marijuana
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Research Foundation for Mental Hygiene, Inc. (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB# 5350; DA09236 (Other Grant/Funding Number: National Institute on Drug Abuse (NIDA))
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Results first posted 2017-12-19 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-02

CONDITIONS: Marijuana Use
Keywords: Naltrexone; Smoked Marijuana
MeSH Terms: conditions — Marijuana Use | interventions — Dronabinol; Naltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blind, placebo-controlled
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (10):
- Placebo, Marijuana (0% THC) (Placebo Comparator): During each session, one capsule containing placebo was administered to the participant in a size 00 opaque capsule with lactose filler. A marijuana cigarette (0% THC; ca. 800 mg) provided by the National Institute on Drug Abuse, was administered 45 minutes post capsule administration.
  Interventions: Drug: Placebo + Inactive Marijuana (0% THC)
- Placebo, Marijuana (3.27% THC) (Experimental): During each session, one capsule containing placebo was administered to the participant in a size 00 opaque capsule with lactose filler. A marijuana cigarette (3.27% THC; ca. 800 mg) provided by the National Institute on Drug Abuse, was administered 45 minutes post capsule administration.
  Interventions: Drug: Placebo + Active Marijuana (3.27% THC)
- Naltrexone (12mg), Marijuana (0% THC) (Experimental): During each session, one capsule containing naltrexone (12 mg) was administered to the participant in a size 00 opaque capsule with lactose filler. A marijuana cigarette (0% THC; ca. 800 mg) provided by the National Institute on Drug Abuse, was administered 45 minutes post capsule administration.
  Interventions: Drug: Naltrexone 12 Mg + Inactive Marijuana (0% THC)
- Naltrexone (12mg), Marijuana (3.27% THC) (Experimental): During each session, one capsule containing naltrexone (12 mg) was administered to the participant in a size 00 opaque capsule with lactose filler. A marijuana cigarette (3.27% THC; ca. 800 mg) provided by the National Institute on Drug Abuse, was administered 45 minutes post capsule administration.
  Interventions: Drug: Naltrexone 12 Mg+ Active Marijuana (3.27% THC)
- Naltrexone (25mg), Marijuana (0% THC) (Experimental): During each session, one capsule containing naltrexone (25 mg) was administered to the participant in a size 00 opaque capsule with lactose filler. A marijuana cigarette (0% THC; ca. 800 mg) provided by the National Institute on Drug Abuse, was administered 45 minutes post capsule administration.
  Interventions: Drug: Naltrexone 25 Mg + Inactive Marijuana (0% THC)
- Naltrexone (25mg), Marijuana (3.27% THC) (Experimental): During each session, one capsule containing naltrexone (25 mg) was administered to the participant in a size 00 opaque capsule with lactose filler. A marijuana cigarette (3.27% THC; ca. 800 mg) provided by the National Institute on Drug Abuse, was administered 45 minutes post capsule administration.
  Interventions: Drug: Naltrexone 25 Mg + Active Marijuana (3.27% THC)
- Naltrexone (50mg), Marijuana (0% THC) (Experimental): During each session, one capsule containing naltrexone (50 mg) was administered to the participant in a size 00 opaque capsule with lactose filler. A marijuana cigarette (0% THC; ca. 800 mg) provided by the National Institute on Drug Abuse, was administered 45 minutes post capsule administration.
  Interventions: Drug: Naltrexone 50 Mg + Inactive Marijuana (0% THC)
- Naltrexone (50mg), Marijuana (3.27% THC) (Experimental): During each session, one capsule containing naltrexone (50 mg) was administered to the participant in a size 00 opaque capsule with lactose filler. A marijuana cigarette (3.27% THC; ca. 800 mg) provided by the National Institute on Drug Abuse, was administered 45 minutes post capsule administration.
  Interventions: Drug: Naltrexone 50 Mg+ Active Marijuana (3.27% THC)
- Naltrexone (100mg), Marijuana (0% THC) (Experimental): During each session, one capsule containing naltrexone (100 mg) was administered to the participant in a size 00 opaque capsule with lactose filler. A marijuana cigarette (0% THC; ca. 800 mg) provided by the National Institute on Drug Abuse, was administered 45 minutes post capsule administration.
  Interventions: Drug: Naltrexone 100 Mg + Inactive Marijuana (0% THC)
- Naltrexone (100mg), Marijuana (3.27% THC) (Experimental): During each session, one capsule containing naltrexone (100 mg) was administered to the participant in a size 00 opaque capsule with lactose filler. A marijuana cigarette (3.27% THC; ca. 800 mg) provided by the National Institute on Drug Abuse, was administered 45 minutes post capsule administration.
  Interventions: Drug: Naltrexone 100 Mg+ Active Marijuana (3.27% THC)

INTERVENTIONS:
Drug: Placebo + Inactive Marijuana (0% THC) — One capsule containing placebo was administered to the participant in a size 00 opaque capsules with lactose filler 45 minutes before marijuana administration.
  Other Names: treatment type 1
  Arms: Placebo, Marijuana (0% THC)
Drug: Placebo + Active Marijuana (3.27% THC) — One capsule containing placebo was administered to the participant in a size 00 opaque capsules with lactose filler 45 minutes before administration of a marijuana cigarette containing 3.27% THC (ca. 800 mg) provided by the National Institute on Drug Abuse.
  Other Names: treatment type 2
  Arms: Placebo, Marijuana (3.27% THC)
Drug: Naltrexone 12 Mg+ Active Marijuana (3.27% THC) — One capsule containing 12mg Naltrexone was administered to the participant in a size 00 opaque capsules with lactose filler 45 minutes before active marijuana administration.
  Other Names: Treatment type 3
  Arms: Naltrexone (12mg), Marijuana (3.27% THC)
Drug: Naltrexone 25 Mg + Active Marijuana (3.27% THC) — One capsule containing 12mg Naltrexone was administered to the participant in a size 00 opaque capsules with lactose filler 45 minutes before active marijuana administration.
  Other Names: treatment type 4
  Arms: Naltrexone (25mg), Marijuana (3.27% THC)
Drug: Naltrexone 50 Mg+ Active Marijuana (3.27% THC) — One capsule containing 25mg Naltrexone was administered to the participant in a size 00 opaque capsules with lactose filler 45 minutes before marijuana administration.
  Other Names: treatment type 5
  Arms: Naltrexone (50mg), Marijuana (3.27% THC)
Drug: Naltrexone 100 Mg+ Active Marijuana (3.27% THC) — One capsule containing 50mg Naltrexone was administered to the participant in a size 00 opaque capsules with lactose filler 45 minutes before marijuana administration.
  Other Names: treatment type 6
  Arms: Naltrexone (100mg), Marijuana (3.27% THC)
Drug: Naltrexone 12 Mg + Inactive Marijuana (0% THC) — One capsule containing 12mg Naltrexone was administered to the participant in a size 00 opaque capsules with lactose filler 45 minutes before inactive marijuana administration.
  Other Names: treatment type 7
  Arms: Naltrexone (12mg), Marijuana (0% THC)
Drug: Naltrexone 25 Mg + Inactive Marijuana (0% THC) — One capsule containing 25mg Naltrexone was administered to the participant in a size 00 opaque capsules with lactose filler 45 minutes before inactive marijuana administration.
  Other Names: treatment type 8
  Arms: Naltrexone (25mg), Marijuana (0% THC)
Drug: Naltrexone 50 Mg + Inactive Marijuana (0% THC) — One capsule containing 50mg Naltrexone was administered to the participant in a size 00 opaque capsules with lactose filler 45 minutes before inactive marijuana administration.
  Other Names: treatment type 9
  Arms: Naltrexone (50mg), Marijuana (0% THC)
Drug: Naltrexone 100 Mg + Inactive Marijuana (0% THC) — One capsule containing 100mg Naltrexone was administered to the participant in a size 00 opaque capsules with lactose filler 45 minutes before inactive marijuana administration.
  Other Names: treatment type 10
  Arms: Naltrexone (100mg), Marijuana (0% THC)

SUMMARY:
The purpose of this study is to determine if the subjective effects of marijuana will be decreased by low-doses (< 25 mg) of naltrexone and increased by high-doses (> 50 mg) of naltrexone.

DETAILED DESCRIPTION:
Laboratory animal studies demonstrate that endogenous cannabinoids and opioids are closely inter-related. We have completed a series of studies in marijuana smokers showing that a clinically-utilized dose of naltrexone (50 mg) enhanced the reinforcing and subjective effects of orally-administered tetrahydrocannabinol (THC), while a low naltrexone dose (12 mg) blunted the effects of THC. A better understanding of the effects of a range of naltrexone doses in combination with smoked marijuana has important implications for the following reasons: (1) Alcohol- and opioid-dependent patients receive high doses of naltrexone (50-150 mg), which may increase the abuse liability of marijuana, (2) Low-dose naltrexone blunts THC's intoxicating effects, suggesting potential utility as a treatment medication for marijuana dependence. This study will determine if naltrexone (0, 12, 25, 50, 100 mg) administration 45 min prior to marijuana administration (0, 3.27% THC) alters marijuana's subjective, cognitive or physiological effects. Marijuana smokers will spend approximately 5h/day for a total of 10 days in the outpatient laboratory. Participants will visit the outpatient laboratory 2-3 times per week, with a minimum 48-hr interval between sessions to allow for naltrexone clearance. These data will provide important information regarding the clinical use of naltrexone.

ELIGIBILITY:
Inclusion Criteria:

* Current marijuana use
* Able to perform study procedures
* 21-45 years of age
* Women practicing an effective form of birth control

Exclusion Criteria:

* Current, repeated illicit drug use (other than marijuana)
* Presence of significant medical illness (e.g., diabetes, cardiovascular disease, hypertension, examination, laboratory hepatitis, clinically significant laboratory abnormalities, tests, 12-lead ECG, Mantoux test LFTs > 3x upper limit of normal)
* History of heart disease
* Request for drug treatment
* Current parole or probation
* Pregnancy or current lactation
* Recent history of significant violent behavior
* Previous adverse reaction to naltrexone
* Major current Axis I psychopathology Psychiatric interview (e.g., major depressive disorder, bipolar disorder, suicide risk, schizophrenia)
* Current use of any prescription or over-the-counter medication

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2006-12; Primary Completion 2008-05 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Haney, Ph.D., Principal Investigator — New York State Psychiatric Institute

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 15 males and 14 females completed this study, which used a within-subject design such that each participant received 10 different drug treatments/interventions in total.
Groups:
- Overall Study Participant Flow: Of the 49 participants enrolled, only 29 completed all 10 drug interventions.
Period: Overall Study
Arm/Group | Overall Study Participant Flow
Started | 49
Completed | 29
Not Completed | 20

BASELINE CHARACTERISTICS:
Groups:
- Overall Number of Baseline Participants: Baseline measures are only reported for the 29 participants who completed the study.
Arm/Group | Overall Number of Baseline Participants
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.0 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Subjective Mood Scores as a Function of Marijuana Strength and Naltrexone Dose.
Description: All subjective effects were measured using visual analog scales (VAS), a series of 100 mm long lines labeled 'not at all' at one end (0 mm) and 'extremely' at the other end (100 mm). Participants were instructed to rate their subjective experiences on the line according to how they felt at that particular moment. Subjective assessments included measures of perceived marijuana strength, marijuana "high", "good effects" of marijuana, and how much marijuana was "liked".
  Marijuana's effects were determined by comparing the active and inactive marijuana conditions when paired with the placebo naltrexone condition (one comparison). Naltrexone's intrinsic effects were assessed by comparing placebo and each active dose of naltrexone (12, 25, 50, and 100 mg) under the inactive marijuana condition (four comparisons). Finally, the active marijuana- placebo naltrexone condition was compared to the active marijuana-active naltrexone conditions (four comparisons)
Time Frame: Baseline compared to 6 week timepoint
Population: Data from 29 participants were included in this analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo + Marijuana (0.0%THC): Placebo + Marijuana (0.0%THC)
- Placebo + Marijuana (3.27% THC): Placebo + Marijuana (3.27% THC)
- Naltrexone (12mg) + Marijuana (0.0%THC): Naltrexone (12mg) + marijuana (0.0%THC)
- Naltrexone (12mg) + Marijuana (3.27%THC): Naltrexone (12mg) + marijuana (3.27%THC)
- Naltrexone (25mg) + Marijuana (0.0%THC): Naltrexone (25mg) + marijuana (0.0%THC)
- Naltrexone (25mg) + Marijuana (3.27%THC): Naltrexone (25mg) + marijuana (3.27%THC)
- Naltrexone (50mg) + Marijuana (0.0%THC): Naltrexone (50mg) + marijuana (0.0%THC)
- Naltrexone (50mg) + Marijuana (3.27%THC): Naltrexone (50mg) + marijuana (3.27%THC)
- Naltrexone (100mg) + Marijuana (0.0%THC): Naltrexone (100mg) + marijuana (0.0%THC)
- Naltrexone (100mg) + Marijuana (3.27%THC): naltrexone + active marijuana
Arm/Group | Placebo + Marijuana (0.0%THC) | Placebo + Marijuana (3.27% THC) | Naltrexone (12mg) + Marijuana (0.0%THC) | Naltrexone (12mg) + Marijuana (3.27%THC) | Naltrexone (25mg) + Marijuana (0.0%THC) | Naltrexone (25mg) + Marijuana (3.27%THC) | Naltrexone (50mg) + Marijuana (0.0%THC) | Naltrexone (50mg) + Marijuana (3.27%THC) | Naltrexone (100mg) + Marijuana (0.0%THC) | Naltrexone (100mg) + Marijuana (3.27%THC)
Number analyzed (Participants) | 29 | 29 | 29 | 29 | 29 | 29 | 29 | 29 | 29 | 29
units on a scale
  Mean VAS ratings "Marijuana Strength" | 8.0 (0.8) | 25.0 (3.2) | 6.7 (0.9) | 34.0 (2.1) | 8.1 (0.6) | 31.6 (1.1) | 9.7 (0.7) | 36.2 (2.3) | 10.1 (0.9) | 34.5 (1.4)
  Mean VAS ratings "High" | 4.1 (0.7) | 11.0 (1.1) | 3.7 (0.6) | 23.0 (3.2) | 3.0 (0.6) | 20.4 (2.2) | 4.0 (0.3) | 22.2 (1.7) | 3.9 (0.3) | 21.3 (2.4)
  Mean VAS ratings "Good Effect" | 10.0 (1.1) | 38.3 (4.5) | 6.8 (1.2) | 43.1 (5.7) | 9.0 (0.8) | 44.1 (5.0) | 10.2 (1.1) | 42.2 (4.2) | 12.5 (0.9) | 44.0 (4.8)
  Mean VAS ratings "Like Drug" | 11.3 (1.2) | 35.0 (5.3) | 7.0 (0.7) | 44.0 (3.7) | 9.3 (1.2) | 34.7 (4.8) | 10.3 (0.5) | 38.0 (6.6) | 11.4 (1.2) | 44.0 (6.0)

2. Primary Outcome: Change in Mean Psychomotor Task Performance as a Function of Marijuana Strength and Naltrexone Dose
Description: Change in Digit Symbol Substitution Test (DSST) scores. Increasing scores indicate improvement, on a scale of 0-90.
  The task batteries included total correct attempts on a 3-min DSST.
Time Frame: Baseline compared to 6 week timepoint
Population: Data from 29 participants were included in this analysis
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Placebo + Marijuana (0.0%THC): Placebo Inactive marijuana (0.0% THC)
  Naltrexone: During each session, one capsule containing placebo or naltrexone (12, 25, 50, and 100 mg) was administered to the participant in a size 00 opaque capsules with lactose filler, prepared by the New York State Psychiatric Institute Research Pharmacy. A marijuana cigarette (0 or 3.27% THC; ca. 800 mg) provided by the National Institute on Drug Abuse was smoked 45 min after naltrexone administration, the time at which naltrexone levels peak.
  Marijuana: During each session, one capsule containing placebo or naltrexone (12, 25, 50, and 100 mg) was administered to the participant in a size 00 opaque capsules with lactose filler, prepared by the New York State Psychiatric Institute Research Pharmacy. A marijuana cigarette (0 or 3.27% THC; ca. 800 mg) provided by the National Institute on Drug Abuse was smoked 45 min after naltrexone administration, the time at which naltrexone levels peak.
- Placebo + Marijuana (3.27% THC): Placebo marijuana (3.27% THC)
  Naltrexone: During each session, one capsule containing placebo or naltrexone (12, 25, 50, and 100 mg) was administered to the participant in a size 00 opaque capsules with lactose filler, prepared by the New York State Psychiatric Institute Research Pharmacy. A marijuana cigarette (0 or 3.27% THC; ca. 800 mg) provided by the National Institute on Drug Abuse was smoked 45 min after naltrexone administration, the time at which naltrexone levels peak.
  Marijuana: During each session, one capsule containing placebo or naltrexone (12, 25, 50, and 100 mg) was administered to the participant in a size 00 opaque capsules with lactose filler, prepared by the New York State Psychiatric Institute Research Pharmacy. A marijuana cigarette (0 or 3.27% THC; ca. 800 mg) provided by the National Institute on Drug Abuse was smoked 45 min after naltrexone administration, the time at which naltrexone levels peak.
- Naltrexone (12mg) + Marijuana (0.0%THC); Naltrexone (25mg) + Marijuana (0.0%THC); Naltrexone (50mg) + Marijuana (0.0%THC); Naltrexone (100mg) + Marijuana (0.0%THC): Naltrexone + Inactive marijuana
- Naltrexone (12mg) + Marijuana (3.27%THC); Naltrexone (25mg) + Marijuana (3.27%THC); Naltrexone (50mg) + Marijuana (3.27%THC); Naltrexone (100mg) + Marijuana (3.27%THC): naltrexone + active marijuana
Arm/Group | Placebo + Marijuana (0.0%THC) | Placebo + Marijuana (3.27% THC) | Naltrexone (12mg) + Marijuana (0.0%THC) | Naltrexone (12mg) + Marijuana (3.27%THC) | Naltrexone (25mg) + Marijuana (0.0%THC) | Naltrexone (25mg) + Marijuana (3.27%THC) | Naltrexone (50mg) + Marijuana (0.0%THC) | Naltrexone (50mg) + Marijuana (3.27%THC) | Naltrexone (100mg) + Marijuana (0.0%THC) | Naltrexone (100mg) + Marijuana (3.27%THC)
Number analyzed (Participants) | 29 | 29 | 29 | 29 | 29 | 29 | 29 | 29 | 29 | 29
units on a scale | 86.2 (1.8) | 86.1 (1.7) | 86.7 (1.7) | 84.7 (1.6) | 83.4 (1.7) | 83.5 (1.6) | 83.6 (1.8) | 82.1 (1.4) | 82.1 (1.6) | 83.0 (1.7)

3. Primary Outcome: Change in Mean Heart Rate as a Function of Marijuana Strength and Naltrexone Dose.
Description: Change in mean heart rate as a function of marijuana and naltrexone dose
Time Frame: Baseline compared to 6 week timepoint
Population: A total of 29 participants were included in the final analysis
Measure: Mean (Standard Deviation); unit: Heart rate (beats/minute)
Arm/Group | Placebo + Marijuana (0.0%THC) | Placebo + Marijuana (3.27% THC) | Naltrexone (12mg) + Marijuana (0.0%THC) | Naltrexone (12mg) + Marijuana (3.27%THC) | Naltrexone (25mg) + Marijuana (0.0%THC) | Naltrexone (25mg) + Marijuana (3.27%THC) | Naltrexone (50mg) + Marijuana (0.0%THC) | Naltrexone (50mg) + Marijuana (3.27%THC) | Naltrexone (100mg) + Marijuana (0.0%THC) | Naltrexone (100mg) + Marijuana (3.27%THC)
Number analyzed (Participants) | 29 | 29 | 29 | 29 | 29 | 29 | 29 | 29 | 29 | 29
Heart rate (beats/minute) | 68.5 (0.5) | 70.7 (0.6) | 65.8 (0.5) | 72.1 (0.4) | 67.3 (0.4) | 72.7 (0.7) | 65.6 (0.3) | 72.2 (0.6) | 67.7 (0.4) | 72.4 (0.4)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the six weeks that each participant was enrolled in the study.
Groups:
- Placebo + Inactive Marijuana (0.0%THC): In this arm, participants received placebo + inactive marijuana (0.0%THC)
- Placebo + Marijuana (3.27% THC): In this arm, participants received placebo + Marijuana (3.27% THC)
- Naltrexone (12mg) + Marijuana (0.0%THC): In this arm, participants received naltrexone (12mg) + marijuana (0.0%THC)
- Naltrexone (12mg) + Marijuana (3.27%THC): In this arm, participants received naltrexone (12mg) + marijuana (3.27%THC)
- Naltrexone (25mg) + Marijuana (0.0%THC): In this arm, participants received naltrexone (25mg) + marijuana (0.0%THC)
- Naltrexone (25mg) + Marijuana (3.27%THC): In this arm, participants received naltrexone (25mg) + marijuana (3.27%THC)
- Naltrexone (50mg) + Marijuana (0.0%THC): In this arm, participants received naltrexone (50mg) + marijuana (0.0%THC)
- Naltrexone (50mg) + Marijuana (3.27%THC): In this arm, participants received naltrexone (50mg) + marijuana (3.27%THC)
- Naltrexone (100mg) + Marijuana (0.0%THC): In this arm, participants received naltrexone (100mg) + marijuana (0.0%THC)
- Naltrexone (100mg) + Marijuana (3.27%THC): In this arm, participants received naltrexone (100mg) + marijuana (3.27%THC)
Arm/Group | Placebo + Inactive Marijuana (0.0%THC) | Placebo + Marijuana (3.27% THC) | Naltrexone (12mg) + Marijuana (0.0%THC) | Naltrexone (12mg) + Marijuana (3.27%THC) | Naltrexone (25mg) + Marijuana (0.0%THC) | Naltrexone (25mg) + Marijuana (3.27%THC) | Naltrexone (50mg) + Marijuana (0.0%THC) | Naltrexone (50mg) + Marijuana (3.27%THC) | Naltrexone (100mg) + Marijuana (0.0%THC) | Naltrexone (100mg) + Marijuana (3.27%THC)
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49 | 0/49 | 0/49 | 0/49 | 0/49 | 0/49 | 0/49 | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49 | 0/49 | 0/49 | 0/49 | 0/49 | 0/49 | 0/49 | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 0/49 | 0/49 | 0/49 | 7/49 | 12/49 | 1/49 | 0/49 | 0/49 | 0/49 | 0/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo + Inactive Marijuana (0.0%THC) (N=49) | Placebo + Marijuana (3.27% THC) (N=49) | Naltrexone (12mg) + Marijuana (0.0%THC) (N=49) | Naltrexone (12mg) + Marijuana (3.27%THC) (N=49) | Naltrexone (25mg) + Marijuana (0.0%THC) (N=49) | Naltrexone (25mg) + Marijuana (3.27%THC) (N=49) | Naltrexone (50mg) + Marijuana (0.0%THC) (N=49) | Naltrexone (50mg) + Marijuana (3.27%THC) (N=49) | Naltrexone (100mg) + Marijuana (0.0%THC) (N=49) | Naltrexone (100mg) + Marijuana (3.27%THC) (N=49)
gastrointestinal upset (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
conflicting social circumstance (Social circumstances) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
A limitation of this study is the small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No